CLINICAL TRIAL: NCT01587287
Title: A Comprehensive Assessment of the Precision and Agreement of Anterior Corneal Power Measurements Obtained Using Different Devices
Brief Title: A Comprehensive Assessment of Anterior Corneal Power by Different Devices
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yifan Feng, Study Director, Wenzhou Medical University
Other Study IDs: YNKT201101
Record Dates: First submitted 2012-04-23; First posted 2012-04-30 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2011-01

CONDITIONS: Myopia
Keywords: Anterior corneal power; Placido topographer; Scheimpﬂug; Precision; Agreement
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Corneal power measurement: All recruited volunteers in present study, that underwent corneal power measurement with 8 different instruments
  Interventions: Device: Corneal power measurement

INTERVENTIONS:
Device: Corneal power measurement — All subjects will be underwent a full ophthalmic examination including vision, auto- and subjective refraction, slit-lamp examination, non-contact tonometry, corneal power measurements with the 8 devices and fundus examination.
  Other Names: Tomey RC-5000

SUMMARY:
To comprehensively assess the precision and agreement of anterior corneal power measurements using 8 different devices.

DETAILED DESCRIPTION:
Volunteers with healthy corneas will be measured by different instruments to detect their anterior corneal power. Only the right eye of each subject was selected. Measurements were repeated in the second session scheduled 1 to 2 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* healthy cornea,
* best corrected distance visual acuity (BCVA) equal to or better than 20/25,
* willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* History of refractive surgery or any keratoplasty procedure,
* use of contact lenses,
* history of corneal dystrophies or degenerative diseases,
* history of glaucoma or ocular hypertension,
* significant subjective dry eye symptoms, Schirmer I test results of less than 5.0 mm, tear film break-up time shorter than 5 seconds and corneal fluorescein staining positive.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The present study's definitions of reproducibility, repeatability and agreement were based on those adopted by the British Standards Institute and the International Organization for Standardization.
  Corneal curvature measurement provides crucial information for calculating intraocular lens power,screening and managing corneal refractive surgeries and corneal disease.
  Volunteers with healthy corneas will be measured by different instruments to detect their anterior corneal power.Only the right eye of each subject was selected.Measurements were repeated in the second session scheduled 1 to 2 weeks later, at almost the same time as the first session, by the same examiner using the same protocol.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Flat corneal power | 2 weeks
  The intrasession repeatability and intersession reproducibility of ﬂat corneal curvature measurements by using the 8 commercially available instruments.
Steep corneal power | 2 weeks
  The intrasession repeatability and intersession reproducibility of Steep corneal curvature measurements by using the 8 commercially available instruments.

SECONDARY OUTCOMES:
Vector power J0 | 2 weeks
  The intrasession repeatability and intersession reproducibility of vector power J0 measurements by using the 8 commercially available instruments.
Vector power J45 | 2 weeks
  The intrasession repeatability and intersession reproducibility of vector power J45 measurements by using the 8 commercially available instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Yifang Feng, MD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Wang Q, Savini G, Hoffer KJ, Xu Z, Feng Y, Wen D, Hua Y, Yang F, Pan C, Huang J. A comprehensive assessment of the precision and agreement of anterior corneal power measurements obtained using 8 different devices. PLoS One. 2012;7(9):e45607. doi: 10.1371/journal.pone.0045607. Epub 2012 Sep 25. PMID 23049823